CLINICAL TRIAL: NCT04156919
Title: Playful Gameplay Broadens Thought-Action Repertoires: Effects of Playfulness on Meaningful Engagement in Health Games
Brief Title: The Impact of a Health Video Game on User-Game Engagement and Dietary Choices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oteng Ntsweng (Other)
Collaborators: Tati Siding Primary School (Unknown); FriendsLearn (Industry)
Responsible Party: Sponsor-Investigator, Oteng Ntsweng, Principal Investigator, National University of Singapore
Organization: National University of Singapore (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Botswana_RCT1
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Dietary Habits; Nutrition Knowledge
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Playful condition (Experimental): Children in the playful and non-playful conditions will receive the fooya! intervention but will be varied in the psychological state of playfulness. Children in the playful condition will play a health game called fooya! Drawing on the playfulness literature, we will manipulate four dimensions of play. First, to manipulate the voluntariness of tasks, children in the playful condition will be asked/invited to participate in the study. Second, to manipulate adult presence, there will be little to no teacher involvement in the playful condition. Third, to manipulate the timing of the activity, children in the playful condition will be given an option to play anytime, including after school hours. Fourth, to manipulate the goal perception, the children in the playful condition will be told that their activity is not graded-i.e., autotelic.
  Interventions: Behavioral: fooya!™
- Non-playful condition (Experimental): As mentioned earlier, we will manipulate four dimensions of play. First, participation will be mandatory for children in the non-playful condition. Second, teacher presence will be more salient in this condition. Third, children in the non-playful condition will participate during school hours. Fourth, the children in the non-playful condition will be told that their activity is graded.
  Interventions: Behavioral: fooya!™
- Control condition (Active Comparator): Children in the control condition will play a video game unrelated to diet and lifestyle called Wordsearch.
  Interventions: Other: WordSearch

INTERVENTIONS:
Behavioral: fooya!™ — fooya!™ is a science/evidence-based AI-enabled neuromodulation and Cognitive Behavior Therapy (CBT) technology. fooya!™ has been shown to deliver statistically significant outcomes concerning food choices during randomized-controlled clinical trials conducted at the Baylor College of Medicine's Children's Nutrition Research in the United States of America as well as India. In the game, children make several decisions with split-second timing, such as food choices, destroying bad/unhealthy food robots using the bad foods that are thrown at the player, and saving themselves. If the children collect good/healthy foods, they are in fit-zone for a while, which shields them from bad food robots.
  Arms: Non-playful condition; Playful condition
Other: WordSearch — We will have an active control group that will play a WordSearch game. The intention is to have the children play a familiar video game through the same modality (IPAD) that is unrelated to diet or lifestyle choices.
  Arms: Control condition

SUMMARY:
Pediatric obesity is one of the most serious public health challenges of the 21st century. It is a serious problem that is expected to create lifelong health challenges and potentially overwhelm the ability of healthcare providers to manage the consequences. While many factors contribute to pediatric obesity, dietary choices are the leading cause. A key concern is how to inculcate healthy dietary habits early among young children. Over the past 20 years, there has been significant scientific interest in examining the potential learning consequences of playing video games given children's interests in such games. This study investigates the impact of a health video game on children's nutritional knowledge and dietary choices.

DETAILED DESCRIPTION:
Brief Overview of the Study Protocol

Study Design, Participants and Recruitment

A cluster randomized controlled trial with three data collection periods-baseline, post one, and post two- will be adopted for this study. We will collaborate with a primary school in the North-East District of Botswana. Recruitment will be done with the help of the school with which we are collaborating. The children will be sent home with consent forms to obtain parental consent. Before participation, eligible parents will provide informed consent and child assent. To ensure sufficient power of 0.8 with a medium effect size, 120 participants will be recruited to participate in the experiment.

Procedures

Following baseline assessment, the children will be randomly assigned to one of three groups: playfulness condition, non-playfulness condition, and control condition. The playfulness and non-playfulness conditions will vary in terms of the climate such that children in the playfulness condition will have a relaxed, play-oriented context while those in the non-playfulness condition will have a more formal work-oriented context. The children in the control condition will play a video game that is unrelated to diet and lifestyle choices. Randomization will be done at the class/cluster level to avoid contamination between the experimental conditions (Puffer et al. 2005). The baseline survey, including demographics and family environment, gaming experience/ frequency of gameplay, nutrition knowledge, social cognitive factors (i.e., attitude, intention, and health locus of control), will be administered after obtaining consent. Since the administration of a pre-test survey may change the way that participants interact with the game (during the experiment) and/or suggest to the participants that there is a socially desirable way to respond to outcome measures, the pre-test survey will be administered a week before the actual experiment. Post 1 experiment data collection will occur immediately upon completion of the experiment. The study will be conducted from November 2019 to May 2020. Post 2 experiment data collection will occur three months after the experiments.

Experimental Setup

Taking into account the malleability of the engagement construct (Boekaerts 2016), we ensured that our setup does not use invasive equipment. The chosen setup thus results from a trade-off between sensitivity and practical requirements. We will use the Tobii pro nano eye tracker that captures gaze data at 60Hz. Skin conductance will be measured using the shimmer 3 GSR kit. It was selected because of its small size and lightweight (28g).

All the experiments will be conducted individually as follows. The participants will sit in a non-swiveling chair in front of an IPAD with an eye tracker. An eye tracker will be attached to the IPAD. The experimenter will begin the session by describing the procedure to the participant. The experimenter will then place physiological feedback sensors to measure skin conductance on the participants' non-dominant hand. The non-dominant hand will be chosen to allow participants free access to the video game touch screen with the dominant hand (Jensen et al. 2016). The participant will be given 6 minutes to feel comfortable, and, at that time, any necessary technical adjustments will be made. We will exclude children who report that they are not comfortable and/or depict symptoms of discomfort. After the participant is comfortable, a survey will be administered to capture their mood. Next, the experimenter will record baseline GSR and gaze data for 2 minutes. To initiate the calibration process for eye gaze data, participants will be required to trace an on-screen object with their eyes (Jensen et al. 2016). Participants will play eight levels of the mobile health game. Based on our pre-tests, the completion of eight levels should take about 20 minutes. This duration was chosen because to prevent myopia, children are advised not to play with handheld devices for more than 30 minutes at a stretch.

After the game, a post-test questionnaire will be administered to capture 1) nutritional knowledge acquisition, 2) subjective emotional responses, 3) social cognitive factors, and 4) perceived game complexity. After completing the post hoc survey, participants will choose four actual food items under the pretext of a parting gift. The following instruction will be used: "thank you for your time. You may now pick what you like from these options. You can eat your choice now or later. It is entirely up to you." The choice will serve as an objective measure of on-site behavior. Following the experiments, we will conduct a follow-up data collection after three months.

ELIGIBILITY:
Inclusion Criteria:

* children in primary level 4 between the ages of 8-11
* children fluent in English
* children who have a parent fluent in English who is willing to participate in the study

Exclusion Criteria:

* children with a history of photosensitive epilepsy
* children with implantable medical devices such as cardiac pacemakers and implantable cardioverter-defibrillators
* underweight children

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Dietary Choice | 1 day
  After each experiment, participants will be asked to choose between six actual food items under the pretext of a parting gift. Of these six, three will be healthy: orange, apple and banana, and three will be unhealthy: potato chips, biscuits and master pop juice. Following prior literature, the gift selection will serve as the onsite objective measure of behavior. We will make sure that the choices are a single small serving so as not to contribute to the problem of unhealthy dietary habits.
Objective Nutrition Knowledge (ONK) | 1 day
  ONK will be captured using the children's identification of healthy foods measure (Tatlow-Golden et al. 2013). Correct answers will be summed to create this formative measure.
Subjective Nutrition Knowledge (SNK) | 1 day
  The SNK measure will be adapted from prior research (Moorman et al. 2004). SNK will be will be assessed using three items: 1) I am able to understand product information on food labels; 2) I know the difference between healthy snacks and unhealthy snacks; 3) I know the difference between healthy drinks and unhealthy drinks. Response options will range from 1=totally disagree to 5=totally agree.
Subjective Experiences of Discrete Emotions | 1 day
  To capture subjective discrete emotions, we will adopt the child version of the positive and negative affect scale, the PANAS-C (Laurent et al. 1999). We select emotions that are relevant to our context (Liu et al. 2017). We will capture six discrete emotions. Of the six, three are positive (excited, joyful, and energetic), and three are negative (upset, nervous, and gloomy).

SECONDARY OUTCOMES:
Health locus of control | 1 day
  health locus of control will be measured by four items, such as "What I eat affects whether I get sick or stay healthy.." Response options will range from 1=totally disagree to 5=totally agree (Genugten et al. 2014).
Dietary Intention | 1 day
  Dietary intake intention will be assessed with one item preceded by the stem: "I plan to..." derived from (Spook et al. 2016). Response options will range from 1=definitely not to 5=definitely.

CONTACTS AND LOCATIONS:
Locations (1):
- Tati Siding Primary School, Tati Siding, North-East District, Botswana

IPD SHARING:
Plan to Share IPD: No